CLINICAL TRIAL: NCT04696393
Title: A Phase 1, Open-Label, Randomized, Two-Period, Crossover Study to Compare the Pharmacokinetics and Safety of Mitapivat 100 mg Tablet Formulation With Mitapivat 2 × 50 mg Tablet Formulation in Healthy Adult Subjects
Brief Title: A Study to Compare the Pharmacokinetics and Safety of Mitapivat 100 mg Tablet Formulation With Mitapivat 2 × 50 mg Tablet Formulation in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-021
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1: AB (Experimental): Participants will receive Treatment A (mitapivat 100 milligram [mg] tablet formulation, orally, under fasted conditions once on Day 1 of Period 1), followed by Treatment B (mitapivat 2 x 50 mg tablet formulation, orally, under fasted conditions once on Day 1 of Period 2). Each treatment period will be separated by a washout period of at least 7 days.
  Interventions: Drug: Mitapivat tablet
- Treatment Sequence 1: BA (Experimental): Participants will receive Treatment B (mitapivat 2 x 50 mg tablet formulation, orally, under fasted conditions once on Day 1 of Period 1), followed by Treatment A (mitapivat 100 mg tablet formulation, orally, under fasted conditions once on Day 1 of Period 2). Each treatment period will be separated by a washout period of at least 7 days.
  Interventions: Drug: Mitapivat tablet

INTERVENTIONS:
Drug: Mitapivat tablet — Oral tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
The primary purpose of this study is to characterize and compare the pharmacokinetic profiles of mitapivat following a single dose administration of 100 mg mitapivat in two tablet formulations (50 mg and 100 mg tablet strengths) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Has the ability to understand the requirements of the study and a willingness to comply with all study procedures and has provided written informed consent before any study-related procedures are conducted, and is willing to comply with all study procedures for the duration of the study;
* Has a body mass index (BMI) ≥18 and ≤32 kilograms per square meter (kg/m^2), at screening;
* Has a body weight ≥50 kg at screening;
* Is medically healthy, with no clinically significant conditions or abnormalities, as determined by the investigator or designee, through evaluation of medical history and vital sign measurements, 12-lead ECG results, physical examination findings, and clinical laboratory test results (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in;
* If female:

  * Is of childbearing potential and agrees to either abstain from sexual intercourse with a male partner or agrees to use a highly effective form of contraception, beginning at screening and continuing throughout the study and for 28 days after dosing or is postmenopausal (defined as 12 months or more continuously with no menses), or
  * Has a documented medical history of tubal ligation or hysterectomy;
  * The following are considered highly effective forms of contraception: hormonal oral contraceptives, injectables, and patches; intrauterine devices; double barrier methods (synthetic condom, diaphragm, or cervical cap used with spermicidal foam, cream, or gel); and male partner sterilization;
* If male (even if vasectomized):

  * Agrees to either abstain from sexual intercourse with a female partner, or
  * Agrees to use a highly effective form of contraception (as defined above), starting at screening and continuing until 90 days after the final dose of mitapivat, and
  * Agrees to not donate sperm throughout the entirety of the study until 90 days after the final dose of mitapivat;
* Agrees to abstain from any alcohol consumption, starting 72 hours prior to check-in and continuing until the follow-up telephone call;
* Agrees to refrain from marijuana- or cannabinol-containing products for 7 days prior to screening until after the follow-up telephone call.

Exclusion Criteria:

* At screening, presents with a condition or has a medical history that, in the opinion of the investigator, may potentially interfere with study drug absorption, distribution, metabolism, and/or excretion (eg, malabsorption [including due to cystic fibrosis, lactose intolerance, celiac disease]);
* At screening, presents with a surgical history that, in the opinion of the investigator, may potentially interfere with study drug absorption, distribution, metabolism, and/or excretion (eg, cholecystectomy). Participants who have undergone abdominal surgery or any other major surgical procedure within 6 months prior to screening, must not be enrolled;
* Has a history or a presence of a primary malignancy, with the exception of a malignancy that has been curatively treated and for which the participant has displayed no evidence of disease within 12 months prior to screening;
* Has a known history or presence of liver disease;
* Is pregnant or breastfeeding;
* Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening;
* Has liver test results including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin that are above the upper limit of normal at screening or check-in (out-of-range test results may be repeated once at screening and check-in, if needed);
* Has estimated glomerular filtration rate (eGFR) <60 milliliters per minute (mL/min)/1.73 m^2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2009 equation;
* Has platelet, hemoglobin, or hematocrit test results that are below the lower limit of normal at screening or check-in (out-of-range test results may be repeated once at screening and check-in, if needed);
* Has confirmed (ie, 2 consecutive measurements) systolic blood pressure (BP) >150 or <90 millimeters of mercury (mmHg), diastolic blood pressure (BP) >90 or <50 mmHg, and pulse rate >100 or <45 beats per minute (bpm) at screening and check-in;
* Has clinically significant cardiac history or presence of ECG findings as determined by the investigator at screening and check-in, including any of the following:

  * Abnormal sinus rhythm (heart rate [HR] lower than 45 bpm and higher than 100 bpm);
  * Risk factors for torsades de pointes (eg, heart failure, cardiomyopathy, or family history of long QT syndrome);
  * Sick sinus syndrome, second- or third-degree atrioventricular block myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities;
  * QT interval corrected for HR using Fridericia's formula (QTcF) >450 milliseconds (msec) (male participants) or >450 msec (female participants). In the event a QTcF value is outside of the reference range, it will be confirmed by 2 further repeat measurements, which will then be used to calculate a mean from the original value and the 2 repeat measurements;
  * QRS interval >110 msec, confirmed by manual over read;
  * PR interval <120 and >220 msec;
  * Repeated or frequent syncope or vasovagal episodes;
  * Hypertension, angina, bradycardia (if assessed as clinically significant by the investigator), or severe peripheral arterial circulatory disorders;
* Has clinically significant laboratory assessment findings, including hypokalemia, hypercalcemia, or hypomagnesemia;
* Has an active infection requiring systemic antimicrobial therapy at any time during the screening period;
* Has a positive urine drug screen (including cotinine) at screening or check-in;
* Has a positive alcohol breath test result or positive urine drug screen at screening or check-in;
* Uses or intends to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including any over-the-counter medications or herbal or nutritional supplements with the exception of vitamins, within 14 days (or 5 half-lives, whichever is longer) prior to check-in and until the follow-up telephone call, unless deemed acceptable by the investigator (or designee). Note: After first dosing, acetaminophen (up to 2 grams per 24 hours) may be administered at the discretion of the investigator or designee;
* Has used any prescription (excluding hormone replacement therapy and hormonal birth control) medications, including systemic antimicrobial therapies, within 30 days (or 5 half-lives, whichever is longer) before the first dose of study drug or during the study (ie, through the follow-up telephone call);
* Is currently enrolled in or has participated in another clinical study to receive any investigational or marketed product or placebo within 2 months (or 5 half-lives, whichever is longer) prior to check-in;
* Has donated blood or blood products or experienced blood loss of >450 mL within 30 days prior to check-in;
* Has received blood products within 2 months prior to check-in;
* Has consumed caffeine- or xanthine-containing products within 24 hours prior to first dose of study drug until after the follow-up telephone call;
* Has consumed foods or beverages containing grapefruit or Seville oranges for 7 days prior to the first dosing and is not willing to refrain from consumption of these foods or beverages throughout the study;
* Has ingested poppy seeds within 7 days prior to check-in until after the follow-up telephone call;
* Has consumed vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussel sprouts, and mustard greens), or charbroiled meats within 7 days prior to first dose of study drug or throughout the study;
* Has used nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, vaporizers, or inhalers) within 6 months prior to screening, based on participant self-reporting, and does not agree to abstain from use until the follow-up telephone call;
* Has a history of active alcoholism or drug/chemical abuse within 2 years prior to check-in;
* Average alcohol consumption of >21 units per week for males and >14 units for females (1 unit is equal to approximately 1/2 pint [200 mL] of beer, or 1 small glass [100 mL] of wine, or 1 measure [25 mL] of 40% spirits);
* Has a history of relevant drug and/or food allergies (ie, allergy to study drug or excipients [microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, magnesium stearate, and mannitol]);
* Has veins that are unsuitable for multiple venipunctures/cannulation, as assessed by the investigator or designee at screening;
* Is involved in strenuous activity or contact sports within 24 hours prior to check-in or throughout the study;
* Has any medical, hematological, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the investigator, may confer an unacceptable risk to participating in the study and/or could confound the interpretation of the study data;
* Has a positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). Note: Testing will be performed according to site procedures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve (AUC) of Mitapivat From Time 0 to the Last Quantifiable Concentration (AUC0-t) | Pre-dose and multiple time points post-dose (up to 120 hours)
AUC of Mitapivat From Time 0 Extrapolated to Infinity (AUC0-inf) | Pre-dose and multiple time points post-dose (up to 120 hours)
Maximum Observed Plasma Concentration (Cmax) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)
Time to Maximum Observed Plasma Concentration (Tmax) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)
Apparent Terminal Elimination Rate Constant (λZ) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)
Terminal Phase Half-life (t1/2) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)
Apparent Oral Clearance (CL/F) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)
Apparent Volume of Distribution (Vd/F) of Mitapivat | Pre-dose and multiple time points post-dose (up to 120 hours)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to approximately 18 days
Number of Participants With Clinically Significant Abnormal Clinical Laboratory Values | Up to approximately 18 days
Number of Participants With Clinically Significant Abnormal Findings for Vital Sign Parameters | Up to approximately 18 days
Number of Participants With Clinically Significant Abnormal Findings for 12-lead Electrocardiogram (ECG) Parameters | Up to approximately 18 days
Number of Participants With Clinically Significant Abnormal Physical Examination Findings | Up to approximately 18 days

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No